CLINICAL TRIAL: NCT06657807
Title: Online Cognitive Behavior Therapy for Anxiety Related to Pediatric Asthma: A Feasibility Study
Brief Title: Online Cognitive Behavior Therapy for Anxiety Related to Pediatric Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marianne Bonnert, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPM Dnr: 2023-01304-01
Record Dates: First submitted 2024-10-03; First posted 2024-10-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Asthma; Anxiety
Keywords: Internet-CBT; Adolescent; Children; Parents
MeSH Terms: conditions — Asthma; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Uncontrolled feasibility study using pretest-posttest design with 2 mo FU as primiary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-CBT (Experimental): Internet-CBT including 8 weekly modules
  Interventions: Behavioral: Online CBT

INTERVENTIONS:
Behavioral: Online CBT — Online CBT targeting anxiety in pediatric asthma
  Other Names: Internet-CBT; Internet-delivered cognitive behavior therapy

SUMMARY:
Asthma is a chronic condition affecting approximately 5-15% of all Swedish children. Research has shown that asthma may be associated with increased anxiety and worry, with children who have asthma being twice as likely to experience anxiety compared to those without asthma. The coexistence of anxiety and asthma can worsen asthma symptoms and heighten anxiety, as it can be challenging to distinguish between the two conditions. Cognitive behavioral therapy (CBT) is a recommended treatment for anxiety in children, but few studies have examined the effectiveness of CBT in children with both asthma and anxiety. Our research group has previously developed internet-delivered CBT (Internet-CBT) targeting anxiety in asthma for adults, yielding promising results. Internet-CBT can significantly improve access to treatment and has been shown to be both effective and safe for other medical conditions.

The primary aim of this project is to investigate whether Internet-CBT can contribute to improved quality of life, better asthma control, and reduced anxiety in children and adolescents whose asthma is complicated by their own or their parents' anxiety. We have previously developed Internet-CBT for adults with asthma and anxiety with promising outcomes. For this study, we have adapted the treatment for children, adolescents, and their parents and will evaluate its feasibility and clinical effectiveness.

DETAILED DESCRIPTION:
This study will use an uncontrolled pretest-posttest design, all participants will receive the intervention. The intervention consists of 8 weekly modules delivered over internet with guided support from an experienced CBT-trained psychologist.

Assessments will be made pretreatment, weekly during treatment for the primary outcome and potential mediators, posttreatment, at the primary endpoint 2 months after treatment completion and at follow up 6 months after treatment completion. Thirty participants (aged 8-17 years) will be included. All outcome data will be collected digitally and include for feasibility: treatment credibility, working alliance, compliance with the treatment (number of modules completed) and with asthma medications as prescribed by the child´s physician, any adverse events, subjective overall relief and satisfaction with treatment. For potential efficacy, the clinical effect in the group will be analyzed on pre- to post-measurements, including weekly measurements and 2 months follow up after treatment termination (primary endpoint). The participants will be followed 6 months after treatment completion to analyze longer term clinical effects.

Recruitment and inclusion procedure Participants will be self-recruited through advertisements in social media and posters at pediatric health care clinics. Potential participants will undergo an online self-report screening of eligible criteria. The parents and adolescents 15 and older, will receive digital information about the study and leave their written consent online. The screening will be followed by an evaluation with a clinical psychologist using a structured interview based on the DSM diagnostic (MINI-KID). During the clinical interview, the children (>age 15) will receive information about the study and leave their informed consent orally. The families will have the opportunity to ask questions about the study and confirm previous written consent.

After inclusion, participants may start their treatment immediately.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years
* A diagnosis of asthma made by a physician and confirmed by the parents
* Some anxiety related to asthma reported by either parent of child ("Do you feel stressed or worried about your asthma?" yes/no) and/or some restriction by asthma in daily life, which could indicate a pattern of avoidance behavior ("Do you feel hindered by your asthma in your daily life?" yes/no)

Exclusion Criteria:

* Presence of severe psychiatric disorders such as severe depression or suicidal ideation.
* Concurrent psychological treatment
* Presence of severe somatic disorder that could interfere with participation in the CBT-treatment
* Other respiratory disease than asthma
* Psychotropic medication should be stable for at least 1 month before entering the study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PedsQL Asthma Module | From pretreatment to 16 weeks
  Questionnarie about asthma symptoms. Participants report how much of a problem asthma have been for them the past month on a scale ranging from 0 (never) to 5 (almost always).

SECONDARY OUTCOMES:
PedsQL Quality of Life Inventory | From pretreatment to 16 weeks
  Questionnaire about Quality of Life. Participants report how much of a problem they/their child has with psychical, emotional, social and study functioning for them the past month on a scale ranging from 0 (never) to 5 (almost always).
Asthma Control Test | From pretreatment to 16 weeks
  Asthma Severity
Asthma Behavior Checklist | From pretreatment to 16 weeks
  Avoidance behavior due to fear of asthma
Fear of Asthma Symptoms Scale | From pretreatment to 16 weeks
  Fear of bodily symptoms of Asthma. Questionnaire where the scale ranges from 0 (never) to 5 (always). A higher score means worse outcome.
Youth Asthma Related Anxiety Scale | From pretreatment to 16 weeks
  Anxiety related to asthma. Questionnaire where the scale ranges from 0 (never) to 5 (always). A higher score means worse outcome.
Subjective Adequate Relief Questionnaire | Week 8
  Subjective Adequate Relief Questionnaire measures self-perceived change in symptoms as a result of the treatment. The scale consists of 2 items rated from 0 (much worse) to 6 (much better).
Client Satisfaction Questionnaire | Week 8
Working Alliance Inventory | Week 3
  Questionnaire used to assess perceived alliance with the online therapist. The questions are scored on a scale from 1 (never) to 7 (always). A higher score means better outcome.
Credibility Rating Scale | Week 2
  The Credibility Scale was developed to assess the participant's expectations of the treatment. The scale ranges from 0 (not at all) to 10 (very much). A higher score means better outcome.
Adverse events | Week 8
Spence Children's Anxiety Scale | From pretreatment to 16 weeks
  Spence Children's Anxiety Scale is used to assess symptoms of anxiety and is specifically developed for children. The scale ranges from never (0) to always (3). A higher score means worse outcome.
Child Depression Inventory | From pretreatment to 16 weeks
Adult responses to children's symptoms | From pretreatment to 16 weeks
  Questionnaire used to assess how parents respond to their children when they have symptoms. The questions are scored on a scale from 0 (never) to 4 (always). A higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Psychiatry Research, Karolinska Institutet & Stockholm Health Care, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided